CLINICAL TRIAL: NCT05247008
Title: Effectiveness of Thyme Honey in Management of Xerostomia in Geriatric Patients With ESRD: Longitudinal Prospective Clinical Biochemical Study
Brief Title: Effectiveness of Thyme Honey in Management of Xerostomia in ESRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 972
Record Dates: First submitted 2021-10-29; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-02

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: Treatment protocol:
  * Thyme honey will topically be applied to the oral mucosa as oral rinse based on the Biswal et al. (2003) administration protocol.
  * Based on this protocol, patients will have oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day.
  * Patients will be instructed to perform thyme honey rinses in the oral mucosa.
  * Patients will be instructed not to swallow the thyme honey oral rinse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thyme honey interventional arm in geriatric patients having end-stage renal disease. (Other): Thyme honey used as mouth rinse in treatment of xerostomia in geriatric patients with end-stage renal disease.
  Interventions: Other: Thyme honey

INTERVENTIONS:
Other: Thyme honey — * Thyme honey will topically be applied to the oral mucosa as oral rinse based on the Biswal et al. (2003) administration protocol.
  * Based on this protocol, patients will have oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day.

SUMMARY:
The oral health of older people has warranted considerable research attention in the last two to three decades. One of the most oral conditions that have been related to the elderly patients was xerostomia.

An elderly population that has a high rate of comorbid disease is likely to continue for the foreseeable future. Among these pathologies, End stage renal disease (ESRD) stands out as a common serious age-related disease. ESRD is a chronic irreversible renal failure. It is known also as chronic kidney disease (CKD) Stage 6 or CKD 6. Xerostomia is relatively common in patients having ESRD with prevalence ranging from 28% to 67%.

Multiple pharmacological and non-pharmacological measures that have been tested in previous studies in order to improve xerostomia in patients with ESRD which were based on the stimulation of the salivary gland flow.

A new alternative for the control of xerostomia is the use of thyme honey, which is a propolis gel product with strong antioxidant, antibacterial, antifungal and immunomodulation effect. It is believed that the presence of honey in the oral cavity has a sialagogue effect, stimulating the salivary glands to produce more saliva, due to the high sugar concentration in honey.

The purpose of the study is to determine whether the use of thyme honey as mouth rinse will help in the treatment of xerostomia in geriatric patients with end-stage renal disease (symptom management).

DETAILED DESCRIPTION:
Most patients with end-stage renal disease (ESRD) on hemodialysis (HD) have to maintain a fluid-restricted diet in order to prevent fluid overload between dialysis sessions. . However, compliance to the fluid restriction is also influenced by other factors, such as hormonal derangements, social and psychological changes, thirst and xerostomia.

Xerostomia in ESRD is a multifactorial phenomenon and various mechanisms contribute to its development as direct uremic involvement of salivary glands, atrophy and fibrosis of the salivary glands, chemical inflammation, dehydration, mouth breathing. The other conditions that may cause dry mouth in uremic patients are retrograde parotitis, metabolic abnormalities, use of diuretics and due to inability of kidneys to reabsorb sodium and the resultant polyuria.

Xerostomia, the subjective feeling of oral dryness, is a symptom most frequently accompanied by either decreased salivary flow or an altered composition of saliva. Hyposalivation, on the other hand, is the objective measured reduction in salivary flow rate. Xerostomia is a relatively common complaint, particularly among older people, and can lead to major consequences with regard to the quality of their general and oral health and wellbeing.

Xerostomia has a variety of possible etiological factors; it is generally classified as having primary and secondary causes. Primary causes comprise conditions that directly affect the salivary glands and induce xerostomia like, Sjogren's syndrome, diabetes mellitus type 1 and 2, thyroid disease, adrenal pathology, renal or hepatic diseases, hepatitis C virus infection, and HIV disease.

Secondary causes of xerostomia include the side-effects of radiation therapy or chemotherapy, rheumatoid arthritis, scleroderma, mixed connective tissues diseases, systemic lupus erythematous, graft versus host disease, anorexia, alcohol and smoking and commonly prescribed drugs (>500 medications reportedly cause dry mouth). The most common medications causing hyposalivation are those with anticholinergic activity, sympathomimetics, and benzodiazepines. The risk of xerostomia increases with the synergistic effects of xerogenic medications, multiple medications, higher doses of medication, and the duration of the medication.

Saliva plays an important role in maintaining the physiological homeostasis of the oral cavity. In addition to humidifying the oral tissues, its lubricating properties aid in swallowing and talking, and also prevent damage due to mechanical agents. Saliva contains a variety of electrolytes, peptides, glycoproteins, enzymes, immunoglobulin A, amines, and leucocytes.

Owing to the multiple functions of saliva, hyposalivation leads to speech problems, taste disorders, chewing and swallowing difficulties, ill-fitting dentures and consequently poor qualities of life. Furthermore, hyposalivation results in decreased oral clearance, declined salivary pH and buffering capacity, and reduced immune defenses. These symptoms may increase risks of developing infectious oral diseases such as cervical caries, periodontitis and oral candidiasis.

Among saliva constituents, the nitric oxide (NO) is a biochemical marker that involved in both physiological and pathological processes of the salivary glands. High concentrations of nitrate and nitrite (stable metabolites of NO) in normal saliva may ensure potentially protective effects, such as antibacterial properties, increased mucosal blood flow, and oral mucus production.

Multiple pharmacological and non-pharmacological measures that have been tested in previous studies in order to improve xerostomia in patients with ESRD which were based on the stimulation of the salivary gland flow. Salivary glands can be stimulated to produce saliva mechanically (for example, by chewing gum, using different formulated mouthwashes or acupressure) or through medications (such as pilocarpine, cevimeline, angiotensin-converting enzyme inhibitors and angiotensin-receptor antagonists.

Overall, the available interventions do not appear to provide an effective, comprehensive and long-term management of xerostomia. This has strengthened the need for further investigation of other interventions for the management of xerostomia.

A new alternative for the control of xerostomia is the use of thyme honey, which is a propolis gel product with strong antioxidant, antibacterial, antifungal and immunomodulation effect. It is believed that the presence of honey in the oral cavity has a sialagogue effect, stimulating the salivary glands to produce more saliva, due to the high sugar concentration in honey.

Honey has been used historically for its medicinal properties. It has been used to heal burns, surgical wounds, and oral infections because of its antibacterial and analgesic agents and epithelialization boosting effect. Honey has no side effects like other pharmaceutical drugs due to its properties.

As Egypt is considered a low-income country, therefore, the general properties of ideal saliva substitutes to be used should be inexpensive, edible, hydrating, safe-to-swallow but retainable in the mouth.

Given the importance of the oral health status of older people with ESRD associated with xerostomia and thinking that the saliva substitutes or stimulants could potentially be used to decrease this complaint, thus, the urge to drink in hemodialysis patients. This may increase compliance to the fluid-restricted diet and could, subsequently, result in improvement in their quality of life. This study is designed to evaluate the efficiency of different and natural treatment as thyme honey in management of geriatric Egyptian patients with xerostomia and its association to the level of salivary nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, of minimum 61 years.

  * All patients must be clinically diagnosed of ESRD undergoing hemodialysis.
  * Patients on hemodialysis ≥ 3 months (Bots et al., 2005).
  * All patients must have complaint of xerostomia.
  * Objective dry mouth score from ( 2-5).
  * Subjective dry mouth score from (1-4).
  * Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol. Healthy patients.
* Patient with history of any serious illness as malignancy, who undergo kidney transplant.
* Patients with any autoimmune disease.
* Patients with diabetes mellitus (Charalambous et al., 2017).
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both genders with end-stage renal disease
Enrollment: 40 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Changes in subjective dry mouth score | one month
  Changes in subjective dry mouth score [ Time Frame: baseline, 2 weeks and 4 weeks after intervention] The outcome measure (subjective dry mouth score) will be measured before and 2 and 4 weeks after continuous usage of thyme honey mouth rinse (for at least 5 days per week)

SECONDARY OUTCOMES:
Increase in unstimulated Salivary Flow Rate (ml/min) | one month
  Increase in unstimulated Salivary Flow Rate (ml/min) [ Time Frame: baseline, 2 weeks and 4 weeks after intervention ] The outcome measure will be measured before and 2 and 4 weeks after continuous usage of thyme honey mouth rinse (for at least 5 days per week)
Increase in salivary Nitric oxide levels (mmol/L) using clorimetric determination method | one month
  Increase in salivary Nitric oxide levels (mmol/L) using clorimetric determination method [ Time Frame: baseline and 4 weeks after intervention] The outcome measure will be measured before and 4 weeks after continuous usage of thyme honey mouth rinse (for at least 5 days per week).
Changes in objective dry mouth score | one month
  Changes in objective dry mouth score [ Time Frame: baseline, 2 weeks and 4 weeks after intervention] The outcome measure will be measured before and 2 and 4 weeks after continuous usage of thyme honey mouth rinse (for at least 5 days per week)
Changes in salivary Potential of Hydrogen ion (pH) | one month
  Changes in salivary Potential of Hydrogen ion (pH) [ Time Frame: baseline, 2 weeks and 4 weeks after intervention ] The outcome measure will be measured before and 2 and 4 weeks after continuous usage of thyme honey mouth rinse (for at least 5 days per week)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
will not share my raw data

REFERENCES:
- [Background] Afsaneh Abadi P, Koopaie M, Montazeri R. Comparison of salivary nitric oxide and oral health in diabetic patients with and without xerostomia. Diabetes Metab Syndr. 2020 Jan-Feb;14(1):11-15. doi: 10.1016/j.dsx.2019.11.014. Epub 2019 Nov 25. PMID 31809967
- [Background] Alam F, Islam MA, Gan SH, Khalil MI. Honey: a potential therapeutic agent for managing diabetic wounds. Evid Based Complement Alternat Med. 2014;2014:169130. doi: 10.1155/2014/169130. Epub 2014 Oct 15. PMID 25386217
- [Background] Anil S, Vellappally S, Hashem M, Preethanath RS, Patil S, Samaranayake LP. Xerostomia in geriatric patients: a burgeoning global concern. J Investig Clin Dent. 2016 Feb;7(1):5-12. doi: 10.1111/jicd.12120. Epub 2014 Sep 1. PMID 25175324
- [Background] Bardow A, Nyvad B, Nauntofte B. Relationships between medication intake, complaints of dry mouth, salivary flow rate and composition, and the rate of tooth demineralization in situ. Arch Oral Biol. 2001 May;46(5):413-23. doi: 10.1016/s0003-9969(01)00003-6. PMID 11286806
- [Background] Belcher J. Dressings and healing with honey. Br J Nurs. 2014 Mar 27-Apr 9;23(6):S22. doi: 10.12968/bjon.2014.23.Sup6.S22. PMID 24690746
- [Background] Biswal BM, Zakaria A, Ahmad NM. Topical application of honey in the management of radiation mucositis: a preliminary study. Support Care Cancer. 2003 Apr;11(4):242-8. doi: 10.1007/s00520-003-0443-y. Epub 2003 Feb 19. PMID 12673463
- [Background] Bossola M. Xerostomia in patients on chronic hemodialysis: An update. Semin Dial. 2019 Sep;32(5):467-474. doi: 10.1111/sdi.12821. Epub 2019 May 22. PMID 31117154
- [Background] Bots CP, Brand HS, Veerman EC, Valentijn-Benz M, Van Amerongen BM, Valentijn RM, Vos PF, Bijlsma JA, Bezemer PD, Ter Wee PM, Amerongen AV. Interdialytic weight gain in patients on hemodialysis is associated with dry mouth and thirst. Kidney Int. 2004 Oct;66(4):1662-8. doi: 10.1111/j.1523-1755.2004.00933.x. PMID 15458464
- [Background] Bots CP, Brand HS, Veerman EC, Korevaar JC, Valentijn-Benz M, Bezemer PD, Valentijn RM, Vos PF, Bijlsma JA, ter Wee PM, Van Amerongen BM, Nieuw Amerongen AV. Chewing gum and a saliva substitute alleviate thirst and xerostomia in patients on haemodialysis. Nephrol Dial Transplant. 2005 Mar;20(3):578-84. doi: 10.1093/ndt/gfh675. Epub 2005 Jan 21. PMID 15665029
- [Background] Breseghelo Mde L, Guillo LA, Nogueira TE, Leles CR. Nitric Oxide Concentration and Other Salivary Changes after Insertion of New Complete Dentures in Edentulous Subjects. Int J Dent. 2016;2016:8351427. doi: 10.1155/2016/8351427. Epub 2016 Feb 29. PMID 27034674
- [Background] Charalambous A, Lambrinou E, Katodritis N, Vomvas D, Raftopoulos V, Georgiou M, Paikousis L, Charalambous M. The effectiveness of thyme honey for the management of treatment-induced xerostomia in head and neck cancer patients: A feasibility randomized control trial. Eur J Oncol Nurs. 2017 Apr;27:1-8. doi: 10.1016/j.ejon.2017.01.001. Epub 2017 Jan 16. PMID 28279391
- [Background] Cho EP, Hwang SJ, Clovis JB, Lee TY, Paik DI, Hwang YS. Enhancing the quality of life in elderly women through a programme to improve the condition of salivary hypofunction. Gerodontology. 2012 Jun;29(2):e972-80. doi: 10.1111/j.1741-2358.2011.00594.x. Epub 2011 Nov 30. PMID 22126433
- [Background] Dalodom S, Lam-Ubol A, Jeanmaneechotechai S, Takamfoo L, Intachai W, Duangchada K, Hongsachum B, Kanjanatiwat P, Vacharotayangul P, Trachootham D. Influence of oral moisturizing jelly as a saliva substitute for the relief of xerostomia in elderly patients with hypertension and diabetes mellitus. Geriatr Nurs. 2016 Mar-Apr;37(2):101-9. doi: 10.1016/j.gerinurse.2015.10.014. Epub 2015 Nov 26. PMID 26631691
- [Background] Davison SN, Jhangri GS. Impact of pain and symptom burden on the health-related quality of life of hemodialysis patients. J Pain Symptom Manage. 2010 Mar;39(3):477-85. doi: 10.1016/j.jpainsymman.2009.08.008. PMID 20303025
- [Background] Villa A, Wolff A, Aframian D, Vissink A, Ekstrom J, Proctor G, McGowan R, Narayana N, Aliko A, Sia YW, Joshi RK, Jensen SB, Kerr AR, Dawes C, Pedersen AM. World Workshop on Oral Medicine VI: a systematic review of medication-induced salivary gland dysfunction: prevalence, diagnosis, and treatment. Clin Oral Investig. 2015 Sep;19(7):1563-80. doi: 10.1007/s00784-015-1488-2. Epub 2015 May 22. PMID 25994331
- [Background] Vinke J, Kaper HJ, Vissink A, Sharma PK. Dry mouth: saliva substitutes which adsorb and modify existing salivary condition films improve oral lubrication. Clin Oral Investig. 2020 Nov;24(11):4019-4030. doi: 10.1007/s00784-020-03272-x. Epub 2020 Apr 17. PMID 32303864
- [Background] Wolff A, Joshi RK, Ekstrom J, Aframian D, Pedersen AM, Proctor G, Narayana N, Villa A, Sia YW, Aliko A, McGowan R, Kerr AR, Jensen SB, Vissink A, Dawes C. A Guide to Medications Inducing Salivary Gland Dysfunction, Xerostomia, and Subjective Sialorrhea: A Systematic Review Sponsored by the World Workshop on Oral Medicine VI. Drugs R D. 2017 Mar;17(1):1-28. doi: 10.1007/s40268-016-0153-9. PMID 27853957
- [Background] Yang G, Lin S, Wu Y, Zhang S, Wu X, Liu X, Zou C, Lin Q. Auricular Acupressure Helps Alleviate Xerostomia in Maintenance Hemodialysis Patients: A Pilot Study. J Altern Complement Med. 2017 Apr;23(4):278-284. doi: 10.1089/acm.2016.0283. Epub 2017 Feb 13. PMID 28191857
- [Background] Yang LY, Chen HM, Su YC, Chin CC. The effect of transcutaneous electrical nerve stimulation on increasing salivary flow rate in hemodialysis patients. Oral Dis. 2019 Jan;25(1):133-141. doi: 10.1111/odi.12948. Epub 2018 Sep 9. PMID 30076692
- [Background] Yang LY, Yates P, Chin CC, Kao TK. Effect of acupressure on thirst in hemodialysis patients. Kidney Blood Press Res. 2010;33(4):260-5. doi: 10.1159/000317933. Epub 2010 Jul 2. PMID 20606475
- [Background] Yu IC, Tsai YF, Fang JT, Yeh MM, Fang JY, Liu CY. Effects of mouthwash interventions on xerostomia and unstimulated whole saliva flow rate among hemodialysis patients: A randomized controlled study. Int J Nurs Stud. 2016 Nov;63:9-17. doi: 10.1016/j.ijnurstu.2016.08.009. Epub 2016 Aug 20. PMID 27565424
- [Derived] Ibrahim SS, Abou-Bakr A, Ghalwash DM, Hussein RR. Effectiveness of thyme honey in the management of xerostomia in geriatric patients with end-stage renal disease: a randomized controlled clinical trial with a biochemical assessment. Eur J Med Res. 2023 Oct 7;28(1):406. doi: 10.1186/s40001-023-01351-9. PMID 37805605